CLINICAL TRIAL: NCT00384410
Title: Use of the Cannabinoid Nabilone for the Promotion of Sleep in Chronic, Non-Malignant Pain Patients: A Placebo-Controlled, Randomized, Crossover Insomnia Pilot Study
Brief Title: Use of the Cannabinoid Nabilone for the Promotion of Sleep in Chronic, Non-Malignant Pain Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Bausch Health Americas, Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NAB-20051
Record Dates: First submitted 2006-10-04; First posted 2006-10-06 (Estimated); Last update posted 2006-10-06 (Estimated); Status verified 2005-11

CONDITIONS: Pain; Insomnia
Keywords: Pain; Insomnia; Nabilone
MeSH Terms: conditions — Pain; Sleep Initiation and Maintenance Disorders | interventions — nabilone

INTERVENTIONS:
Drug: Nabilone

SUMMARY:
Sleep disturbance is perhaps one of the most prevalent complaints of patients with long-standing painful conditions. Nabilone is a medication that is approved by Health Canada as an anti-emetic (prevent vomiting) for patients undergoing chemotherapy. Nabilone, due to its sleep promoting properties, is sometimes prescribed by physicians to pain patients to help improve their sleep. However, there is no direct research evidence to either support or refute this practice. This study will investigate if nabilone is effective in improving sleep in insomnia and pain patients.

DETAILED DESCRIPTION:
Rationale:

The current evidence suggests a sleep promoting effect of THC. Although, there is some support from pre-clinical and small sample size human studies suggesting a direct sleep enhancing effect, it remains unclear from the larger clinical trials, whether improved sleep is an epiphenomena secondary to improvements in the primary outcome measures ( i.e., pain, nausea or spasticity). There are no studies evaluating the sleep promoting effects of THC or analogues in patients with primary insomnia or objectively evaluating sleep at baseline and following treatment with THC or analogues in patients suffering from chronic pain disorder and insomnia. Cannabinoids have the potential of simultaneously improving sleep and lessening chronic, non-malignant pain, thereby interrupting the vicious cycle of pain and sleep disturbance. An investigation of the efficacy of cannabinoids in treating insomnia in chronic, non-malignant pain patients is therefore warranted.

Research Question:

To evaluate if nabilone (Cesamet) is effective in improving sleep in patients with insomnia and chronic, non-malignant pain

ELIGIBILITY:
Inclusion Criteria

* History of insomnia and chronic, non-malignant pain.
* Patient not currently being prescribed opiates for pain management
* Subject has no known clinically significant abnormal vital signs or other significant clinical findings at screening.

Exclusion criteria

* Patients with a history of sensitivity of cannabinoids.
* Patients currently taking hypnotics, psychotomimetic substances, CNS depressants or tricyclic antidepressants that may increase the CNS-depressant effects of nabilone.
* Patients with active cardiac disease or respiratory disorders.
* Patients with a history of psychotic reactions, schizophrenia, bipolar disorder or any serious untreated mental disorder.
* Presence of untreated sleep disorder (other than insomnia) as detected using the screening overnight PSG.
* Alcohol or substance abuse (according to DSM-IV) during the last 6 months prior to baseline.
* Patients with liver disease that may interfere with the clearance of nabilone.
* Patients who are nursing, pregnant or likely to become pregnant throughout the course of the study. During the study, female patients will be asked to use an effective method of birth control.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16
Dates: Start 2005-12

PRIMARY OUTCOMES:
The primary analysis variable will be the change in the mean of the sleep efficiency as measured by overnight polysomnography.

SECONDARY OUTCOMES:
• The key secondary efficacy variable will be the change in the total sleep time with nabilone treatment as compared to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Colin M. Shapiro, MBBCh, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada